CLINICAL TRIAL: NCT05586880
Title: A Randomized, Placebo-controlled, Double-blind Crossover Study to Evaluate Efficacy of EnXtra on Accuracy & Reaction Time, Perceived Alertness & Digital Fatigue for Video Gamers
Brief Title: Study to Evaluate Efficacy of EnXtra on Accuracy & Reaction Time, Perceived Alertness & Digital Fatigue for Video Gamers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: OM/220502/ENXTRA/RTPADF
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Alert Fatigue, Health Personnel
MeSH Terms: conditions — Alert Fatigue, Health Personnel | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, Crossover Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EnXtra 300 mg/ capsule (Experimental): One capsule to be taken 3±0.5 hours prior to second gaming session on Day 1 followed by 1 capsule daily after breakfast for 5 days
  Interventions: Other: Experimental: EnXtra 300 mg/ capsule
- Microcrystalline cellulose (MCC) 300mg (Placebo Comparator): One capsule to be taken 3±0.5 hours prior to second gaming session on Day 1 followed by 1 capsule daily after breakfast for 5 days
  Interventions: Other: Microcrystalline cellulose (MCC) 300mg

INTERVENTIONS:
Other: Experimental: EnXtra 300 mg/ capsule — One capsule to be taken 3±0.5 hours prior to second gaming session on Day 1 followed by 1 capsule daily after breakfast for 5 days
  Arms: EnXtra 300 mg/ capsule
Other: Microcrystalline cellulose (MCC) 300mg — One capsule to be taken 3±0.5 hours prior to second gaming session on Day 1 followed by 1 capsule daily after breakfast for 5 days
  Arms: Microcrystalline cellulose (MCC) 300mg

SUMMARY:
In the present study, Sponsor aim to evaluate the effects of EnXtra® as to improve Accuracy & Reaction Time, Perceived Alertness & Digital Fatigue for Video Gamers. A Randomized, Placebo-controlled, Double-blind Crossover Study of 60 randomized cross over for total study duration of approximately 25 days with 5 days of treatment period for each arm and 5-7 days wash out period between both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Males & Females aged ≥ 18 - ≤ 40 years.
2. Subjects with Body Mass Index (BMI) 18 - 29.9 kg/ m2
3. Subjects with history of playing video games for 6 or more hours/ week for 6 months before the screening
4. Subject who can read and understand English language with ease.
5. Fasting blood glucose (FBG) ≤ 125 mg/dl
6. Subjects with history of regular sleep and agree to sleep for 8 ±1 hours the night before the visit day.
7. Subjects who agree to maintain their usual dietary habits and level of exercise i.e. maintain their usual life-style throughout the trial period.
8. Subjects willing to refrain from consuming alcohol 24 hours prior to the visit days.
9. Subjects willing to refrain from consuming caffeine and caffeine-containing products 24 hour prior to visit days.
10. Willing to participate in the study with a signed and dated written consent.

Exclusion Criteria:

1. Subjects suffering from Insomnia.
2. Subjects suffering from chronic fatigue, stress or anxiety.
3. Subjects with uncontrolled hypertension with systolic blood pressure ≥130 and diastolic blood pressure ≥89 mm Hg.
4. Subjects with uncontrolled Type II Diabetes Mellitus with FBG >125 mg/ dl
5. Subjects with Hemoglobin (Hb) ≤ and/or ≥ 13.5 - 17.0 g/Dl inmales and 12.0 - 15.0 g/dL in females.
6. Subjects with ≤ and/or ≥ Total Leucocyte Counts (TLC) 4.0 - 10.0 x 10 3/U
7. Subjects with Differential Leukocyte Counts (DLC) outside the normal range. [Neutrophils: 40 - 80 %, Lymphocytes: 20 - 40 %, Monocytes: 2 - 10 %, Eosinophils: 1 - 6 %, Basophils: 0 - 0.02 %]
8. Subjects with AST values ≤ and/or ≥ 40 U/L in males and 32 U/Lin females.
9. Subjects with ALT values ≤ and/or ≥ 41 U/L in males and 33 U/Lin females
10. Subjects with Creatinine ≤ and/or ≥ Males: 59-104 μmol/L in males and 45-84 μmol/L in females
11. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders.
12. Chronic Alcoholics and smokers
13. Subjects taking any medications or preparations to improve gaming performance (herbal, dietary supplements, homeopathic preparations, etc.) and/or cognitive performance during the study.
14. Subjects who have any other disease or condition, or are using any medication, that in the judgment of the investigator may interfere with evaluations in the study or noncompliance with treatment or visits.
15. Subjects who are on anxiolytics, anti-depressants, antipsychotics, anticonvulsants, antihypertensive, centrally acting corticosteroids, opioid pain relievers, hypnotics, and/or prescribed sleep medications.
16. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
17. Subjects who have had participated in a study of an investigational product 90 days prior to the screening.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Reaction Accuracy | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP & 3 hours post IP on Day 5; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & 3 hours post IP on Day 15
  Reaction Accuracy as assessed by change in the accuracy score for the video game (Call of Duty) as compared to the placebo
Reaction Time | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP & 3 hours post IP on Day 5; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & 3 hours post IP on Day 15
  Reaction Time as assessed by change in the time to response using stroop effect as compared to the placebo

SECONDARY OUTCOMES:
TIME | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP & 3 hours post IP on Day 5; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & 3 hours post IP on Day 15
  Time taken to complete the mission for the video game (Call of Duty) as compared to the placebo
Stanford Sleepiness Scale | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP & Day 5 - 3 hours post IP; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & Day 15 - 3 hours post IP
  Perceived Alertness after video game assessed by change in Stanford Sleepiness Scale (SSS) after video game session, as compared to that of placebo
  Higher the score is the worst outcome and lowest the score is the better outcome.
Multidimensional Fatigue Inventory mental domain scores | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP & Day 5 - 3 hours post IP; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & Day 15 - 3 hours post IP
  Mental fatigue as assessed by change in Multidimensional Fatigue Inventory (MFI) mental domain scores at the end of the video game, as compared to the placebo The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. This tool has been tested for its psychometric properties in individuals receiving radiotherapy, those with the chronic fatigue syndrome, psychology students, medical students, army recruits and junior physicians
Multidimensional Fatigue Inventory physical domain scores | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP, Day 5 - 3 hours post IP; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & Day 15 - 3 hours post IP
  Physical fatigue as assessed by change in Multidimensional Fatigue Inventory (MFI) physical domain score at the end of the video game, as compared to the placebo The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. This tool has been tested for its psychometric properties in individuals receiving radiotherapy, those with the chronic fatigue syndrome, psychology students, medical students, army recruits and junior physicians
Multidimensional Fatigue Inventory (MFI) motivation domain scores | Day 1 - Pre - IP (Baseline), Day 1 - 3 hours post IP, Day 5 - 3 hours post IP; Day 10 - Pre - IP (Baseline), Day 10 - 3 hours post IP & Day 15 - 3 hours post IP
  Intrinsic motivation for video gaming as assessed by change in the Multidimensional Fatigue Inventory (MFI) motivation domain scores after game session, as compared to placebo.
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. This tool has been tested for its psychometric properties in individuals receiving radiotherapy, those with the chronic fatigue syndrome, psychology students, medical students, army recruits and junior physicians

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Principal Investigator — Vedic Lifesciences Pvt. Ltd.
Locations (2):
- India (2):
  - Dr D Y Patil medical college, Nerul, Maharashtra
  - Dr. Sarala Kataria Clinic, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: No